CLINICAL TRIAL: NCT00987467
Title: Long-term Results of Topical Cyclosporine 0.05% in the Treatment of Atopic Keratoconjunctivitis
Brief Title: Long-term Topical Cyclosporine for Atopic Keratoconjunctivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00010864
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Results first posted 2013-10-08 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Atopic Keratoconjunctivitis
Keywords: Atopic; Keratoconjunctivitis; Restasis; Cyclosporine
MeSH Terms: conditions — Keratoconjunctivitis | interventions — Cyclosporine; Vision, Ocular; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyclosporine 0.05% ophthalmic (Experimental): cyclosporine 0.05% ophthalmic eye drops will be used starting with 1 drop in both eyes 6 times daily for first month, followed by 1 drop in both eyes 4 times daily for the following month, then will be adjusted by clinician as needed for appropriate disease control
  Interventions: Drug: Cyclosporin 0.05% ophthalmic

INTERVENTIONS:
Drug: Cyclosporin 0.05% ophthalmic — Cyclosporine 0.05% ophthalmic solution, 1 drop 6 times in both eyes daily for first month, then 1 drop 4 times in both eyes daily for next month, then dosage was adjusted based on clinical disease by investigator.
  Other Names: Restasis

SUMMARY:
Atopic keratoconjunctivitis (AKC) is a rare type of ocular allergy that is often associated with eczema. Over time, the complications from this disease process lead to loss of vision due to continual scarring of the corneal surface. The pathophysiology of AKC has not been fully elucidated, and the triggers are still unknown.

Corticosteroids are very effective in controlling the acute symptoms of AKC. However, two thirds of patients managed with a combination of oral antihistamine, topical mast cell stabilizer, and intermittent topical steroid regimen eventually developed significant keratopathy and vision loss. Additionally, there are many side effects of corticosteroids, including local immunosuppression, cataract formation, and increased risk of glaucoma.

Cyclosporin A is an immunomodulator that specifically inhibits T lymphocytes by blocking the expression of the interleukin-2 receptor. It also blocks the release of inflammatory mediators from mast cells and eosinophils. Cyclosporin has no known side effects except for burning upon instillation, and safe to use over long-term . The investigators have demonstrated that a 0.05% ophthalmic emulsion of cyclosporine has been shown to be effective at improving the ocular signs and symptoms of AKC over short-term. However, the long-term efficacy of cyclosporine A in slowing the natural history of AKC and possible steroid sparing effects have not been assessed. The investigators hypothesize that cyclosporine A can be used as a mainstay treatment of AKC to control signs and symptoms over a long period of time and also prevent the progression of this disease.

DETAILED DESCRIPTION:
Atopic keratoconjunctivitis (AKC) is a rare type of ocular allergy that is often associated with eczema. Over time, the complications from this disease process lead to loss of vision due to continual scarring of the corneal surface. The pathophysiology of AKC has not been fully elucidated, and the triggers are still unknown.

Corticosteroids are very effective in controlling the acute symptoms of AKC. However, two thirds of patients managed with a combination of oral antihistamine, topical mast cell stabilizer, and intermittent topical steroid regimen eventually developed significant keratopathy and vision loss. Additionally, there are many side effects of corticosteroids, including local immunosuppression, cataract formation, and increased risk of glaucoma.

Cyclosporin A is an immunomodulator that specifically inhibits T lymphocytes by blocking the expression of the interleukin-2 receptor. It also blocks the release of inflammatory mediators from mast cells and eosinophils. Cyclosporin has no known side effects except for burning upon instillation, and safe to use over long-term . The investigators have demonstrated that a 0.05% ophthalmic emulsion of cyclosporine has been shown to be effective at improving the ocular signs and symptoms of AKC over short-term. However, the long-term efficacy of cyclosporine A in slowing the natural history of AKC and possible steroid sparing effects have not been assessed. The investigators hypothesize that cyclosporine A can be used as a mainstay treatment of AKC to control signs and symptoms over a long period of time and also prevent the progression of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient has known diagnosis of atopic keratoconjunctivitis
* Patient has been on cyclosporine 0.05% eye drops for control of atopic keratoconjunctivitis
* Patient has been followed up for at least for 1 year
* Patient is able to give informed consent
* Patient is able to tolerate a full ophthalmic exam

Exclusion Criteria:

* Patient has any other diagnosis (i.c. vernal keratoconjunctivitis, giant papillary conjunctivitis) that may alter the clinical appearance or behavior of their ocular surface)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esen K Akpek, MD, Principal Investigator — Johns Hopkins Hospital - Wilmer Eye Institute
Locations (1):
- Johns Hopkins Hospital - Wilmer Eye Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Akpek EK, Dart JK, Watson S, Christen W, Dursun D, Yoo S, O'Brien TP, Schein OD, Gottsch JD. A randomized trial of topical cyclosporin 0.05% in topical steroid-resistant atopic keratoconjunctivitis. Ophthalmology. 2004 Mar;111(3):476-82. doi: 10.1016/j.ophtha.2003.05.035. PMID 15019322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the PI's medical clinic.
Pre-assignment Details: Patients started with a conjunctival biopsy prior to enrolling in the study. Following biopsy, for one week, patients were discontinued on antiinflammatories and given only topical antibiotic prior to the study treatment of topical cyclosporin.
Groups:
- Cyclosporine: Patients with atopic keratoconjunctivitis were started with cyclosporine 0.05% ophthalmic eye drops, starting with 1 drop in both eyes 6 times daily for first month, followed by 1 drop in both eyes 4 times daily for the following month, then adjusted by clinician as needed for appropriate disease control.
  Cyclosporins : Cyclosporine 0.05% ophthalmic solution, 6 times in both eyes daily for first month, then 4 times in both eyes daily for next month, then dosage was adjusted based on clinical disease by investigator
Period: Overall Study
Arm/Group | Cyclosporine
Started | 12
Completed | 10
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cyclosporine
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Ocular Symptoms and Signs Total Composite Score
Description: Symptoms (itching, tearing, discomfort, discharge, photophobia) and signs (Bulbar conjunctival hyperemia, upper tarsal conjunctival papillae, punctate keratitis, corneal neovascularization, cicatrizing conjunctivitis, and blepharitis) evaluated on a 4 point scale of 0-3, with a minimum symptom score of 0- maximum 15, and sign score minimum 0- maximum 18. These scores are combined to yeild a total composite score of signs and symptoms of minimum 0-maximum 33. The highest score would indicate the most severe case of Atopic Keratoconjunctivitis (AKC). The composite score is reported.
Time Frame: Baseline and 8 weeks
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Patients With Steroid Resistant/ Dependant AKC.: Ten patients with significant AKC either steroid dependent or resistant who were having active inflammation were enrolled in this study.
Arm/Group | Patients With Steroid Resistant/ Dependant AKC.
Number analyzed (Participants) | 10
units on a scale
  Baseline | 29.1 [14 to 40]
  8 weeks | 4.7 [0 to 15]
Statistical Analysis 1: Comparison: Patients With Steroid Resistant/ Dependant AKC; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Corticosteroid Usage
Description: Number of flare-ups requiring topical steroid-use across all participants over the entire 12 month follow-up period
Time Frame: Entire follow-up period (Approximately 12 months)
Measure: Number; unit: Total number of flare-up episodes
Groups:
- Topical Steroid Resistant/Dependant AKC: Patients with topical steroid resistant or dependant AKC were used for this study.
Arm/Group | Topical Steroid Resistant/Dependant AKC
Number analyzed (Participants) | 10
Total number of flare-up episodes | 3

ADVERSE EVENTS:
Arm/Group | Cyclosporine
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
We were not able to have a control group and the treatment was not masked.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No